CLINICAL TRIAL: NCT04045327
Title: A Prospective, Multi-Centric, Randomized, Double-Blind, Parallel, Phase-III Study to Assess Efficacy of PMZ-2010 as a Resuscitative Agent for Hypovolemic Shock to be Used as an Adjuvant to Standard Shock Treatment
Brief Title: Efficacy of PMZ-2010 (Centhaquine) a Resuscitative Agent for Hypovolemic Shock
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmazz, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PMZ-2010/CT-3.1/2018; CTRI/2019/01/017196 (Registry Identifier: Clinical Trials Registry - India)
Record Dates: First submitted 2019-07-31; First posted 2019-08-05 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Hypovolemic Shock
MeSH Terms: conditions — Shock | interventions — Saline Solution; centhaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Saline (Active Comparator): Hypovolemic shock patients will be provided the standard of care. Following randomization 100 ml (equal volume to experimental arm) of normal saline will be administered intravenously over 1 hour.
  Interventions: Drug: Normal saline + Standard Treatment
- PMZ-2010 (centhaquine) (Experimental): Hypovolemic shock patients will be provided the standard of care. Following randomization PMZ-2010 (0.01 mg/kg) will be administered intravenously over 1 hour in 100 mL of normal saline.
  Interventions: Drug: Centhaquine + Standard Treatment

INTERVENTIONS:
Drug: Normal saline + Standard Treatment — Normal Saline to be Used as Vehicle in the Phase-III Study to Assess Efficacy of PMZ-2010 as a Resuscitative Agent for Hypovolemic Shock
  Other Names: Vehicle
  Arms: Normal Saline
Drug: Centhaquine + Standard Treatment — Phase-III Study to Assess Efficacy of PMZ-2010 as a Resuscitative Agent for Hypovolemic Shock
  Other Names: PMZ-2010
  Arms: PMZ-2010 (centhaquine)

SUMMARY:
This is a prospective, multi-centric, randomized, double-blind, parallel, controlled phase-III efficacy clinical study of PMZ-2010 therapy in patients with hypovolemic shock.

Centhaquine (previously used names, centhaquin and PMZ-2010; International Non-proprietary Name (INN) recently approved by WHO is centhaquine) has been found to be an effective resuscitative agent in rat, rabbit and swine models of hemorrhagic shock, it decreased blood lactate, increased mean arterial pressure, cardiac output, and decreased mortality. An increase in cardiac output during resuscitation is mainly attributed to an increase in stroke volume. Centhaquine acts on the venous α2B-adrenergic receptors and enhances venous return to the heart, in addition, it produces arterial dilatation by acting on central α2A-adrenergic receptors to reduce sympathetic activity and systemic vascular resistance.

DETAILED DESCRIPTION:
Approximately 105 patients will be randomized 2:1 into 2 treatment groups after meeting the eligibility criteria. Total 70 patients will be enrolled in PMZ-2010 group (Group 1) and in Normal Saline group (Group 2) total 35 patients will be enrolled.

* Group 1: PMZ-2010 (Dose: 0.01 mg/kg) + Standard of care
* Group 2: Normal Saline (Dose: Equal volume) + Standard of care In both treatment groups, patients will be provided the standard of care. PMZ-2010 or Normal Saline will be administered intravenously after randomization to hypovolemic shock patients with systolic arterial blood pressure ≤ 90 mmHg at presentation and continue to receive standard Shock Treatment. In PMZ-2010 group, dose of PMZ-2010 (0.01 mg/kg) will be administered as an intravenous (IV) infusion over 1 hour in 100 mL of normal saline. Second dose of PMZ-2010 will be administered if SBP falls below or remains below or equal to 90 mmHg but not before 4 hours of previous dose and total doses per day (in 24 hours) will not exceed 3 doses. PMZ-2010 administration if needed will continue for two days post randomization. Minimum 1 dose or maximum 6 doses of PMZ-2010 will be administered within first 48 hours. post randomization. In Control group, single dose of equal volume of Normal Saline will be administered as intravenous (IV) infusion over 1 hour in 100 mL of normal saline post randomization. Condition of administration will remain same as for PMZ-2010 group. Each patient will be monitored closely throughout his/her hospitalization and will be followed until discharge from randomization. Each patient will be assessed for efficacy parameters over 28 days from randomization to a clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypovolemic shock admitted to the emergency room or ICU with systolic blood pressure ≤ 90 mmHg at presentation and continue to receive standard shock treatment. Blood Lactate level indicative of hypovolemic shock (>2.0 mmol/L).

Exclusion Criteria:

1. Development of any other terminal illness not associated with Hypovolemic shock during the 28-day observation period.
2. Patient with altered consciousness not due to Hypovolemic shock.
3. Known pregnancy.
4. Cardiopulmonary resuscitation (CPR) before randomization.
5. Presence of a do not resuscitate order.
6. Patient is participating in another interventional study.
7. Patients with systemic diseases which were already present before having trauma, such as: cancer, chronic renal failure, liver failure, decompensated heart failure or AIDS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure | 48 hours
  Change in systolic and diastolic blood pressure - Mean through 48 hours
Change in blood lactate level | 48 hours
  Change in blood lactate level - Mean through 48 hours
Change in base-deficit | 48 hours
  Change in Base-deficit - Mean through 48 hours

SECONDARY OUTCOMES:
Total Urine Output | 48 hours
  Total volume of urine output - Mean through 48 hours
Vasopressor(s) infused | 48 hours
  Amount of total vasopressor(s) infused - Mean through 48 hours
Volume of fluid administered | 48 hours
  Total volume of fluid administered - Mean through 48 hours
Doses of study drug | 48 hours
  Number of doses of study drug administered in first 48 hours post randomization
Incidence of mortality | 28 days
  Proportion of patients with all-cause mortality at 48 hours and 28 days
Stay in hospital, in ICU and/or on Ventilator | 28 days
  Days in hospital, in ICU and/or on Ventilator - Mean through 28 days
Change in Multiple Organ Dysfunction Syndrome Score | 28 days
  Change in Multiple Organ Dysfunction Syndrome Score (MODS) - Mean through 28 days. MODS is a 5 grade scale from 0 to 4, where 0 is the best and 4 is the worst outcome.
Change in Acute Respiratory Distress Syndrome | 28 days
  Change in Acute Respiratory Distress Syndrome (ARDS) - Mean through 28 days. ARDS will be determined using Murray Score for Acute Lung Injury which is based upon radiological findings, oxygenation status, ventilation status of the patient. A lower score of 0 is the best and about 2.5 is the worst outcome.
Change in Glasgow coma score | 28 days
  Change in Glasgow coma score (GCS) - Mean through 28 days. GCS is a 15 point scale to assess the level of consciousness of patients where less than 3 is comatose state and 15 is fully awake.
Incidence of adverse events | 28 days
  Proportion of patients with drug related adverse events during 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Anil Gulati, MD, PhD, Study Chair — Pharmazz, Inc.
Locations (18):
- India (18):
  - Seven Star Hospital, Nagpur, Maha
  - Jawahar Lal Nehru Medical College & Attached Hospitals, Ajmer
  - Radiant Superspeciality Hospital, Amravati
  - People Tree Hospitals, Bangalore
  - KLE's Dr. Prabhakar Kore Hospital & Medical Research Centre, Belagavi
  - Shri Guru Ram Rai Institute of Medical & Health Sciences, Dehradun
  - Department of Surgery, GSVM Medical College, Kanpur
  - Institute of Postgraduate Medical Education & Research and SSKM Hospital, Kolkata
  - King George's Medical University, Lucknow
  - Christian Medical College & Hospital, Ludhiana
  - Sidhu Hospital Pvt. Ltd., Ludhiana
  - Department of General Medicine, JSS Hospital, Mysuru
  - New Era Hospital & Research Institute, Nagpur
  - Rahate Surgical Hospital & ICU, Nagpur
  - Criticare Hospital & Research Institute, Nagpur
  - ACSR Government Medical College & Hospital, Nellore
  - Maulana Azad Medical College and associated Lok Nayak Hospital, New Delhi
  - Institute of Medical Sciences, Banaras Hindu University, Varanasi

IPD SHARING:
Plan to Share IPD: No
Plan to publish the findings after completion of the study

REFERENCES:
- [Background] Kontouli Z, Staikou C, Iacovidou N, Mamais I, Kouskouni E, Papalois A, Papapanagiotou P, Gulati A, Chalkias A, Xanthos T. Resuscitation with centhaquin and 6% hydroxyethyl starch 130/0.4 improves survival in a swine model of hemorrhagic shock: a randomized experimental study. Eur J Trauma Emerg Surg. 2019 Dec;45(6):1077-1085. doi: 10.1007/s00068-018-0980-1. Epub 2018 Jul 13. PMID 30006694
- [Background] Papalexopoulou K, Chalkias A, Pliatsika P, Papalois A, Papapanagiotou P, Papadopoulos G, Arnaoutoglou E, Petrou A, Gulati A, Xanthos T. Centhaquin Effects in a Swine Model of Ventricular Fibrillation: Centhaquin and Cardiac Arrest. Heart Lung Circ. 2017 Aug;26(8):856-863. doi: 10.1016/j.hlc.2016.11.008. Epub 2016 Dec 19. PMID 28385449
- [Background] Papapanagiotou P, Xanthos T, Gulati A, Chalkias A, Papalois A, Kontouli Z, Alegakis A, Iacovidou N. Centhaquin improves survival in a swine model of hemorrhagic shock. J Surg Res. 2016 Jan;200(1):227-35. doi: 10.1016/j.jss.2015.06.056. Epub 2015 Jun 29. PMID 26216751
- [Background] Gulati A, Zhang Z, Murphy A, Lavhale MS. Efficacy of centhaquin as a small volume resuscitative agent in severely hemorrhaged rats. Am J Emerg Med. 2013 Sep;31(9):1315-21. doi: 10.1016/j.ajem.2013.05.032. Epub 2013 Jul 19. PMID 23871440
- [Background] Lavhale MS, Havalad S, Gulati A. Resuscitative effect of centhaquin after hemorrhagic shock in rats. J Surg Res. 2013 Jan;179(1):115-24. doi: 10.1016/j.jss.2012.08.042. Epub 2012 Sep 2. PMID 22964270
- [Background] Gulati A, Lavhale MS, Garcia DJ, Havalad S. Centhaquin improves resuscitative effect of hypertonic saline in hemorrhaged rats. J Surg Res. 2012 Nov;178(1):415-23. doi: 10.1016/j.jss.2012.02.005. Epub 2012 Apr 2. PMID 22487389
- [Result] Anil Gulati, Dinesh Jain, Nilesh Agrawal, Prashant Rahate, Soumen Das, Rajat Chowdhuri, Deba Dhibar, Madhav Prabhu, Sameer Haveri, Rohit Agarwal, Manish Lavhale. Clinical Phase II Results Of PMZ-2010 (centhaquin) As A Resuscitative Agent For Hypovolemic Shock. Critical Care Medicine Volume 47, Issue 1, Page 12.
- [Derived] Gulati A, Choudhuri R, Gupta A, Singh S, Ali SKN, Sidhu GK, Haque PD, Rahate P, Bothra AR, Singh GP, Maheshwari S, Jeswani D, Haveri S, Agarwal A, Agrawal NR. A Multicentric, Randomized, Controlled Phase III Study of Centhaquine (Lyfaquin(R)) as a Resuscitative Agent in Hypovolemic Shock Patients. Drugs. 2021 Jun;81(9):1079-1100. doi: 10.1007/s40265-021-01547-5. Epub 2021 Jun 1. PMID 34061314
- [Derived] Gulati A, Choudhuri R, Gupta A, Singh S, Noushad Ali SK, Sidhu GK, Haque PD, Rahate P, Bothra AR, Singh GP, Maheshwari S, Jeswani D, Haveri S, Agarwal A, Agrawal NR. A multicentric, randomized, controlled phase III study of centhaquine (Lyfaquin (R) ) as a resuscitative agent in hypovolemic shock patients. medRxiv [Preprint]. 2021 May 9:2020.07.30.20068114. doi: 10.1101/2020.07.30.20068114. PMID 33173916